CLINICAL TRIAL: NCT03140202
Title: Impact of a Feedback Device, CPRmeter®, on Chest Compression Quality Preservation During Cardio-pulmonary Resuscitation: A Manikin Study
Brief Title: Compression Is Life In Cardiac Arrest - Quality Study (CILICA-QS)
Acronym: CILICA-QS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: A16-D51-VOL.30
Record Dates: First submitted 2017-04-24; First posted 2017-05-04 (Actual); Last update posted 2017-07-19 (Actual); Status verified 2017-04

CONDITIONS: Cardiac Arrest
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Intervention Model Description: In Guide group, participants have a real time feedback (and record) on chest compression quality performed by means of the visuals informations profided by the feedback device.
  In Blind group, participants have a real time record of chest compression quality performed by means of the feedback device without feedback information of the performance.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Guide then blind (Experimental): This group use the CPRmeter visual feedback during cardiopulmonary resuscitation (screen visible) first, then have no access to the CPRmeter visual feedback during cardiopulmonary resuscitation (screen mask).
  Interventions: Device: CPRmeter (feedback device) with feedback; Device: CPRmeter (feedback device) without feedback
- Blind then guide (Experimental): This group have no access to the CPRmeter visual feedback during cardiopulmonary resuscitation (screen mask) first then use the CPRmeter visual feedback during cardiopulmonary resuscitation (screen visible).
  Interventions: Device: CPRmeter (feedback device) with feedback; Device: CPRmeter (feedback device) without feedback

INTERVENTIONS:
Device: CPRmeter (feedback device) with feedback — Participants have a real time feedback and record.
Device: CPRmeter (feedback device) without feedback — Participants have a real time record without feedback.

SUMMARY:
Context: Chest compressions quality is known to be essential in cardiopulmonary resuscitation. Despite a known harmful effect of chest compressions interruptions, current guidelines still recommend provider switch every 2 minutes. Feedback impact on chest compressions quality preservation during cardiopulmonary resuscitation remains to be assessed.

Study design: simulated prospective monocentric randomized crossover trial.

Participants and methods: Sixty five professionals rescuers of the pre-hospital care unit of University Hospital of Caen (doctors, nurses and ambulance drivers) are enrolled to performed continuous chest compression on manikin (ResusciAnne®, Laerdal), twice, with and without a feedback device (CPRmeter®). Correct compression score (the main criterion) is defined by reached target of rate, depth and leaning at the same time (recorded continuously).

Hypothesis: Feedback device preserve chest compression quality above the 2 minutes recommended switch over during cardiopulmonary resuscitation.

ELIGIBILITY:
Inclusion Criteria:

* Operational staff of University hospital of Caen pre-hospital unit
* Ability in CardioPulmonary Resuscitation

Exclusion Criteria:

* medical contraindication
* refusal

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2017-04-18 (Actual); Primary Completion 2017-09-15 (Estimated); Study Completion 2017-10-01 (Estimated)

PRIMARY OUTCOMES:
Correct compression score | Day 0
  Correct compression score is defined by reached target of rate (between 100/min and 120/min), depth (between 50 mm and 60 mm) and leaning (less than 2500g) at the same time

SECONDARY OUTCOMES:
Decrease time of 30% of correct compression score | Day 0
  Time at witch correct compression score decrease of 30% of the reference correct compression score (first 20 secondes)
Chest compression depth | Day 0
  Chest compression depth reached (in mm)
Chest compression rate | Day 0
  Chest compression rate per min
Percentage of chest compression without leaning | Day 0
  Percentage of chest compression without leaning defined with a residual weight egal or above 2500 g
Percentage of chest compression with correct depth | Day 0
  Percentage of chest compression with depth between 50 mm and 60 mm
Percentage of correct chest compression rate | Day 0
  Percentage chest compression rate between 100/min and 120/min
Participants' fatigue (Borg's scale) | Day 0
  Participant auto-evaluation of fatigue with a predefined scale from 6 to 20 (no unit).

OTHER OUTCOMES:
Hemodynamic effect n1 of Cardiopulmonary Resuscitation | Day 0
  Impact of Cardiopulmonary Resuscitation effort on participant blood pressure (mmHg)
Hemodynamic effect n2 of Cardiopulmonary Resuscitation | Day 0
  Impact of Cardiopulmonary Resuscitation effort on participant heart frequency (/min)

CONTACTS AND LOCATIONS:
Overall Officials: Clement BULEON, MD, Principal Investigator — Medical Simulation Center Normandie Simulation en Sante
Locations (1):
- University Hospital of Caen, Caen, Normandy, France

IPD SHARING:
Plan to Share IPD: No